CLINICAL TRIAL: NCT02604628
Title: Community-acquired Pneumonia: Increasing Protocol Adherence by Antibiotic Stewardship in a Stepped Wedge Cluster- Randomized Trial
Brief Title: Increasing Community-acquired Pneumonia Protocol Adherence by Antibiotic Stewardship
Acronym: CAP-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, MJM Bonten, Prof., UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia; Antibiotic Stewardship; Stepped wedge; Antibiotic
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients will be treated as standard of care.
- Antibiotic Stewardship Intervention (Experimental): Patients will be treated as standard of care. The Antibiotic Stewardship Intervention will be targeted at the physicians treating the community-acquired pneumonia patients. The purpose of the intervention is to increase prescription concordance with the national guideline for community-acquired pneumonia.
  Interventions: Behavioral: Antibiotic Stewardship Intervention

INTERVENTIONS:
Behavioral: Antibiotic Stewardship Intervention — The Antibiotic Stewardship Intervention will consist of education, motivating opinion leaders, adapting a pragmatic disease severity classification and prospective audit and feedback.
  Arms: Antibiotic Stewardship Intervention

SUMMARY:
The purpose of this study is to determine the effect of a multifaceted antibiotic stewardship intervention on protocol adherence of moderate-severe community-acquired pneumonia.

DETAILED DESCRIPTION:
The purpose of the study is to show a decrease in broad-spectrum antibiotics with a non-inferiority in 90-day mortality. Hospitals with a pre-intervention protocol adherence of >70% are excluded from the primary analysis. Primary analysis will be done with a mixed effects model with a random effects for clusters and time. Crude outcomes and outcomes adjusted for potential confounders will be reported. Primary analysis will be tested one-sided for a decrease in mortality. Secondary analysis to test two-sided for mortality will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CAP who get admitted to a non-ICU department are eligible for inclusion.

Exclusion Criteria:

* Patients aged below 18 years
* Residence in a nursing home or long-term care facility in the last 14 days
* Patients hospitalized in an acute care hospital for two or more days in the last 14 days
* Patients with a history of Cystic Fibrosis
* Patients with immunodeficiency, defined as having one or more of the following criteria:

  * HIV infection with a last CD4 count of <300//μL
  * Cytotoxic chemotherapy or radiotherapy in the previous 3 months
  * Chronic hemodialysis > 3 months
  * History of receiving an organ or bone marrow transplant
  * Using immunosuppressive therapy, include corticosteroid treatment only when dosage is high (>0,5mg/kg/day) for a longer period of time (>14 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4084 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Broad-spectrum antibiotic use | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Antibiotic use will be registered during hospital stay
90-day mortality | 90-days after hospital admission
  All-cause mortality on day 90 from admission will be assessed from the municipal personal records database

SECONDARY OUTCOMES:
30-day mortality | 30-days after hospital admission
  All-cause mortality on day 30 from admission will be assessed from the municipal personal records database
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 1 week
Clostridium difficile infections | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Clostridium difficile polymerase chain reaction (PCR) outcomes will be registered during hospital stay
Length of intravenous antibiotic treatment | Participants will be followed for the duration of hospital stay, an expected average of 1 week
Complications | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Complications of pneumonia during admission are registered from the clinical record
Hospital readmissions | Hospital readmissions within 30 days of hospital admission will be registered
  Hospital readmissions will be registered 30 days after hospital admission
Antibiotic switches | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Switches from intravenous to oral (and vice versa) and switches from broad-spectrum to narrow-spectrum (and vice versa) will be registered
Intensive Care admissions | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Intensive Care admissions will be registered during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Marc J.M. Bonten, MD, PhD, Principal Investigator — UMC Utrecht
Locations (12):
- Netherlands (12):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Wilhelmina hospital, Assen
  - Amphia hospital, Breda
  - Catharina hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Ziekehuisgroep Twente, Hengelo
  - Tergooi, Hilversum
  - Erasmus MC, Rotterdam
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Langeland hospital, Zoetermeer

REFERENCES:
- [Derived] Schweitzer VA, van Heijl I, Boersma WG, Rozemeijer W, Verduin K, Grootenboers MJ, Sankatsing SUC, van der Bij AK, de Bruijn W, Ammerlaan HSM, Overdevest I, Roorda-van der Vegt JMM, Engel-Dettmers EM, Ayuketah-Ekokobe FE, Haeseker MB, Dorigo-Zetsma JW, van der Linden PD, Boel CHE, Oosterheert JJ, van Werkhoven CH, Bonten MJM; CAP-PACT Study Group. Narrow-spectrum antibiotics for community-acquired pneumonia in Dutch adults (CAP-PACT): a cross-sectional, stepped-wedge, cluster-randomised, non-inferiority, antimicrobial stewardship intervention trial. Lancet Infect Dis. 2022 Feb;22(2):274-283. doi: 10.1016/S1473-3099(21)00255-3. Epub 2021 Oct 7. PMID 34627499

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT02604628/SAP_000.pdf